CLINICAL TRIAL: NCT05884411
Title: Evaluation of Left Bundle Branch Area Pacing As A Rescue Strategy for Cardiac Resynchronization Therapy Non-response in Patients With Heart Failure: A Randomized Controlled Trial
Brief Title: Evaluation of Left Bundle Branch Area Pacing As A Rescue Strategy for Cardiac Resynchronization Therapy Non-Response
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unsuccessful recruitment
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARA-001-22F; CX002525 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2023-04-28; First posted 2023-06-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Systolic Heart Failure; Heart Failure With Reduced Ejection Fraction; CRT Non-Response; Left Bundle Branch Area Pacing
Keywords: Heart Failure; CRT; LBBAP; Non-response; Cardiac MRI; CMR; Left bundle branch area pacing; cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either receive the new pacing lead in the left bundle branch area or continue current cardiac therapy (CRT) with biventricular CRT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LBBAP (Experimental): This arm will investigate improvement in cardiac function following placement of the LBBA pacing electrode in half the patients.
  Interventions: Device: Left bundle branch area pacing
- Cardiac MRI with devices (Experimental): This arm will investigate the feasibility of cardiac MRI to be used to measure cardiac function in patients with cardiac devices.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Device: Left bundle branch area pacing — A cardiac pacing electrode is inserted into the left bundle branch area of the myocardium via a transvenous approach.
  Other Names: LBBAP
  Arms: LBBAP
Diagnostic Test: Cardiac MRI — A diagnostic imaging test using magnetic resonance imaging to evaluate cardiac function.
  Other Names: CMR
  Arms: Cardiac MRI with devices

SUMMARY:
This study aims to investigate whether the investigators can improve heart function in patients with heart failure who have undergone cardiac resynchronization therapy, but have not had an improvement in their heart function at least one year after the procedure. The investigators will evaluate whether placing a new pacing lead (electrode) in a different part of the heart may increase heart function and decrease heart failure symptoms.

DETAILED DESCRIPTION:
Heart failure is one of the leading causes of death, hospitalization and poor quality of life among Veterans. For many Veterans despite receiving maximal medical therapy for heart failure with reduced ejection fraction (HFrEF), their cardiac function and functional capacity markedly decreases and they develop delays and blocks in their intrinsic conduction system (i.e. left bundle branch block). These patients then meet criteria for cardiac resynchronization therapy (CRT), which has been shown to improve cardiac function. However, up to 40% of patients who undergo CRT do not experience the expected improvement in cardiac function or clinical improvement, and this is termed "non-response".

A critical limitation of traditional CRT is that the leads do not directly utilize the heart's intrinsic conduction tissue, called the His-Purkinje system. An extensive web of conduction tissue capable of transmitting the electrical signals all over the ventricles within milliseconds, the His-Purkinje system conducts electrical stimuli much faster than conduction through a usual myocardial cell. The left bundle branch is a component of the His-Purkinje system. As such, electrophysiologic therapies that directly activate the left bundle branch area (LBBAP) have emerged as possible solutions to the problem of non-response to CRT. Although data suggests that in patients with complete LBBB, LBBAP can better optimize electrical synchrony and improve cardiac function compared to traditional bi-ventricular CRT, the efficacy has not been studied in CRT non-responders.

Currently, the most frequently used technique for assessment of the left ventricle is echocardiography because it is widely available. However, several studies have demonstrated that cardiac MRI (CMR) is superior to echocardiography in measuring left ventricle ejection fraction, particularly in terms of interstudy reproducibility. Recent studies have also demonstrated CMR imaging to be safe even in patients with non-MRI-conditional pacemakers and defibrillators. Studies have also observed that patients undergoing MRI with non-MRI-conditional pacemakers or ICDs neither experienced device/lead failure nor were they at increased risk by undergoing MRI. Despite established safety of CMR in patients with cardiac devices, it is not being routinely performed because there are concerns that the devices will cause field inhomogeneity resulting in magnetic susceptibility artifacts and non-diagnostic image quality. However, these concerns are overcome by utilizing contemporary imaging protocols with gradient echo sequences as opposed to standard steady-state free precession. By using these new protocols for CMR in this study, the investigators aim to establish the feasibility of CMR to prospectively assess cardiac function at baseline and during follow-up in patients with cardiac devices (i.e. that the image quality in subjects with implantable devices is adequate and not undermined by image artifact).

ELIGIBILITY:
Inclusion Criteria:

All Veterans in this study will have undergone CRT at least 12 months prior to enrollment and determined to have non-response by all the following criteria:

* Lack of improvement in New York Heart Association (NYHA) class
* Lack of LVEF increase by > 5%
* Lack of decrease in LVESV by > 15%

Exclusion Criteria:

* Unable to understand or provide informed consent
* Unable or unwilling to participate in the protocol or comply with any of its components
* Pregnant women
* Known cancer patients, actively receiving chemotherapy
* Patients unable to pass MRI safety screening (intra-orbital metallic foreign bodies, severe claustrophobia, etc)
* Patients with anatomical difficulties for implanting LBBAP
* Patients with high risk of procedure-related infection
* Immunocompromised patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction by echocardiography | 6 months
  CRT non-response will be evaluated by echocardiography to assess left ventricular ejection fraction (LVEF). LVEF is reported as a percent.

SECONDARY OUTCOMES:
Left ventricular ejection fraction by cardiac MRI | 6 months
  Cardiac MRI (CMR) will also be used to assess left ventricular ejection fraction (LVEF). LVEF is reported as a percent.
Interventricular mechanical delay measurement by 2D speckle-tracking echocardiography | 6 months
  Left ventricular synchrony will be assessed by measuring the interventricular mechanical delay (measured in ms) using 2D speckle-tracking echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Selma D Carlson, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No